CLINICAL TRIAL: NCT07365618
Title: The Impact of Combined Exercise on Lymphedema, Body Composition, Muscle Strength, and Quality of Life in Breast Cancer Survivors
Brief Title: Combined Exercise Effects in Breast Cancer-related Lymphedema
Acronym: LymFit
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Motricidade Humana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LYMFIT_2025
Record Dates: First submitted 2025-09-08; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer-Related Lymphedema
Keywords: Breast Cancer; Exercise; Fluid Shifts; Edema; Bioelectrical Impedance Analysis
MeSH Terms: conditions — Breast Cancer Lymphedema; Breast Neoplasms; Motor Activity; Edema | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will participate in supervised combined exercise sessions. Additionally, participants will engage in monthly educational sessions.
  Interventions: Behavioral: Exercise; Behavioral: Educational Sessions
- Control Group (Active Comparator): The control group will participate in monthly educational sessions.
  Interventions: Behavioral: Educational Sessions

INTERVENTIONS:
Behavioral: Exercise — Participants randomly allocated to the intervention group will engage in a 12-week combined exercise program, supervised by an accredited exercise physiologist. Sessions will comprise an aerobic component and a resistance component. Exercise progression will be individualized based on participants' tolerance.
  Arms: Experimental Group
Behavioral: Educational Sessions — Participants allocated to both intervention and control groups will attend monthly educational sessions on exercise, nutrition, and other essential health-related topics.

SUMMARY:
Breast cancer-related lymphedema (BCRL) is a common and debilitating condition that affects quality of life, mobility, and well-being. While exercise was once thought to worsen symptoms, current evidence suggests it may improve lymphatic function and symptom management. The LymFit project will test a 12-week combined exercise program (aerobic + resistance) in breast cancer survivors with BCRL compared to usual care.

This investigation aims to unravel the effects of a combined exercise program on BCRL management. A 12-week randomized controlled trial will be conducted with two arms: a combined exercise intervention (strength + aerobic training) and a control group. The LymFit project primarily aims to assess the effects of 12 weeks of combined exercise on L-Dex in BCRL patients. Secondary objectives include evaluating exercise's effects on i) ECW:ICW ratio (dilution techniques); ii) Body composition (dual-energy X-ray absorptiometry), handgrip strength (dynamometry), cardiorespiratory fitness, quality of life, arm disability, anxiety, depression (questionnaires), and inflammatory profile (blood analysis). The project also examines acute exercise (pre- to post-session) responses on iii) Lymphedema (L-Dex) and iv) Fluid shifts (ultrasound muscle thickness + PV measurement). By integrating clinical outcomes with mechanistic evaluations, this randomized controlled trial seeks to generate evidence-based recommendations for exercise in BCRL management and improve understanding of lymphatic fluid dynamics in this population.

DETAILED DESCRIPTION:
- Background - Arm lymphedema is a common, debilitating complication following breast cancer treatment, affecting 20-40% of breast cancer survivors. Breast cancer-related lymphedema (BCRL) is characterized by chronic limb swelling resulting from a significant complication caused by axillary lymph node removal and radiotherapy-induced fibrosis. Symptoms include limb swelling, weakness, decreased mobility, pain, and heaviness, significantly impacting quality of life, daily activities, emotional distress, and social isolation.

Exercise has emerged as a promising non-invasive intervention for BCRL management, supported by leading organizations such as the International Society of Lymphology and the American Society of Breast Surgeons. While traditionally viewed as a risk factor for exacerbating the condition, recent research has highlighted its therapeutic benefits. Strength exercise improves lymphatic function and reduces symptom severity through muscle pump and lymphatic vessel contraction. Aerobic exercise also supports lymph flow through blood circulation and respiration, which creates pressure changes in the thoracic-abdominal cavities and compresses and decompresses lymphatic vessels. Despite the isolated benefits of both types of exercise, the combined exercise (aerobic + strength) may yield additional benefits. However, the effects of combined exercise remain unexplored in BCRL patients. Strength exercise is associated with improved lymphatic function and increased muscle strength, e.g., handgrip strength - a vital health parameter. Aerobic exercise has been linked to enhancements in body composition, cardiometabolic health, inflammatory profile, increased quality of life, and reduced symptoms of anxiety and depression. Therefore, it is justified to explore the potential benefits of combined exercise for patients with BCRL. Although assessing lymphedema remains challenging in clinical practice, the lymphedema index (L-Dex), based on bioelectrical impedance spectroscopy (BIS), provides an objective method for detecting BCRL. The device measures extracellular fluid resistance using the L-Dex ratio, which compares dominant and non-dominant arm values. Although a precise method, it has never been tested in a combined exercise intervention.

From a more mechanistic standpoint, it is known that body water compartments, including total body water (TBW), extracellular water (ECW), and Intracellular water (ICW) plays a crucial role in fluid balance and cellular function. In BCRL, disruptions in this balance - particularly an elevated ECW:ICW (E:I) ratio-may reflect swelling and symptom severity. Research with a clinical population (e.g., elderly or patients with heart failure) suggests that a higher appendicular E:I ratio correlates with lower handgrip and mobility, independent of skeletal muscle mass. These findings suggest that interventions to improve the E:I ratio could enhance overall strength and health. Exercise has been previously demonstrated to improve the E:I ratio in older women and was associated with increased muscle strength. Although our research team has investigated these water compartments in athletes, no study has evaluated them via dilution techniques in BCRL patients. Given the importance of fluid dynamics in lymphedema management, examining these parameters-particularly in response to combined exercise-is crucial to advancing current clinical practice. Another vital point is that acute responses to fluid dynamics have received less attention in research, which may provide insights into the effects of exercise on BCRL and corroborate long-term alterations. Although commonly used, circumferences provide little detailed information about fluids. In contrast, ultrasound combined with plasma volume (PV) analysis has been proposed as a novel method to detect fluid shifts in trained men. Combining ultrasound to assess muscle thickness with PV measurement allows conclusions about acute muscle and vascular fluid, offering insights into the body's response to exercise. This could be valuable for understanding acute fluid mechanisms in BCRL.

In summary, despite progress in BCRL management, gaps remain in understanding the effects of combined exercise on lymphedema and body water compartments. Additionally, research on the acute impact of exercise on fluid mechanisms is needed, as these responses have been less explored in this population. The LymFit project primarily aims to assess the effects of 12 weeks of combined exercise on L-Dex in BCRL patients. Secondary objectives include evaluating exercise's effects on i) E:I ratio (dilution techniques); ii) Body composition (dual-energy X-ray absorptiometry), handgrip strength (dynamometry), cardiorespiratory fitness, quality of life, arm disability, anxiety, depression (questionnaires), and inflammatory profile (blood analysis). The project also examines acute exercise (pre- to post-session) responses on iii) Lymphedema (L-Dex) and iv) Fluid shifts (ultrasound muscle thickness + PV measurement).

* Design - This study will be a randomized controlled trial (RCT) involving a usual care group (UG) and an experimental group (EG) during 12 weeks of intervention. No exercise advice will be provided in the UC, whereas the EG will receive the CDT and three one-hour weekly exercise sessions.
* Hypothesis - A 12-week combined exercise program will: a) reduce the L-Dex in BCRL patients; b) enhance the E:I ratio, indicating improved fluid balance; and c) improve body composition, handgrip strength, cardiorespiratory fitness, quality of life, and inflammatory profile.

A session of combined exercise will induce a) acute reductions in L-Dex, b) increases in muscle thickness (via ultrasound), and c) a reduction in PV.

- Intervention - An accredited exercise physiologist will supervise the three sessions of combined exercise (strength and aerobic) per week during the 12-week intervention. The exercise sessions will follow a structured format designed to allow the intervention to be scalable after the study is completed, enabling its implementation in community programs targeting this population. Accordingly, the exercises will be selected to ensure the intervention can be replicated. The exercise sessions will follow a structured format: The participants will start with a low-intensity warm-up and then proceed to 30 minutes of muscular hypertrophy exercise. Subsequently, participants will perform 20 minutes of aerobic exercise using a static bicycle.

The resistance exercises target the torso's upper and lower limb' muscle groups. Resistance will be set at a weight that participants can lift for 10-12 repetitions, corresponding to an intensity of 5-7 ("somewhat hard-hard") on the OMNI-Resistance Exercise Scale during weeks 1-7 and 7-9 ("hard-extremely hard") during weeks 8-12. Resistance will be increased if participants can lift the weight more than 12 times. If the new weight cannot be lifted, the number of repetitions will be increased from 12 to 14, with instructions to attempt an increase in resistance subsequently. The aerobic exercise consists of cycling on a static bicycle. The target heart rate for the aerobic exercise component will be set at 40-60% (moderate intensity) as recommended by the American College of Sports Medicine (ACSM) of each participant's individualized heart rate reserve (HRR), determined by a graded exercise test performed at the baseline assessments. The Borg scale will be utilized as a subjective measure of perceived exertion throughout the strength session, with a target of 11-12, corresponding to 40-59% of HRR. The aerobic training intensity will be monitored using a heart rate monitor (Polar, H10, Finland). The progression will be individualized depending on the participants' tolerance. Exercise sessions will be monitored and recorded to track progression, compliance, and adherence to the intervention.

- Sample - Participants will be recruited through Hospital Santa Maria in Lisbon and the Associação Nacional de Doentes Linfáticos, collaborating institutions with an extensive database of eligible patients.

The sample size was determined using G*Power v3.1.2, with an α of 0.05, a power of 0.8, and an effect size of 0.27. The effect size was calculated for the primary outcome based on arm L-Dex (our primary outcome), reported in previous research with breast cancer survivors. This calculation yielded a required sample size of 48 participants. To account for a potential dropout rate of approximately 20%, as observed in prior research on exercise interventions in cancer survivors (with reported dropout rates ranging from 5.1% to 19.8%), the total sample size was adjusted to 58 participants (29 in each group).

- Statistical analysis - Statistical analysis will be performed using IBM SPSS Statistics version 29, 2021, for Windows (SPSS Inc., an IBM Company, Chicago, IL, USA).

Descriptive statistics will be employed to characterize the study population at baseline, and data will be summarized using mean and standard deviation for continuous variables and frequencies with percentages for categorical variables. Normality will be assessed for both primary and secondary outcomes using the Shapiro-Wilk test. Linear Mixed Models (LMMs) will evaluate group differences and changes over time. LMMs will account for fixed effects (e.g., group, time, and group-by-time interactions) and random effects to model individual variability. Restricted maximum likelihood estimation (REML) will provide unbiased estimates of variance components. An unstructured covariance matrix will be applied unless model fit indices suggest an alternative covariance structure. Post hoc pairwise comparisons will be conducted using Bonferroni correction to adjust for multiple comparisons. Statistical significance will be set at p < 0.05.

- Contingency plan -

A significant challenge for the LymFit project is maintaining participant adherence throughout the 12-week study duration. As mentioned before, research on exercise interventions in cancer survivors reported dropout rates ranging from 5.1% to 19.8%. The investigators performed a meticulous sample size calculation to prevent a 20% dropout. Still, understanding in advance that the frequency of exercise sessions and assessments may lead to scheduling conflicts, risking reduced compliance, the investigators will address these issues, implementing specific strategies supported by the scientific literature:

1. Expanded recruitment channels: The investigators have multiple recruitment channels, each providing access to a diverse database of potential participants. However, if the recruitment flow proves insufficient, a team member (HSC) maintains professional connections with various hospitals, which can be contacted throughout the study.
2. Capacity to adapt to confounding variables: While the investigators aim to include patients receiving conservative treatments like lymphatic drainage and offer free sessions to standardize access, variability in availability and adherence is expected. If homogenization is unfeasible, our team will leverage its expertise to address this variable in the statistical analysis.
3. Flexible planning: The intervention will last 12 weeks. However, as a contingency measure, the investigators have allocated 8 months to account for potential setbacks. Additionally, the investigators will organize the sample into two cohorts to facilitate the study's management. Participants will also be allowed to attend the FMH facilities at their convenience to receive the intervention, with a team member available to conduct the training rather than adhering to fixed session times.
4. Regular Communication and Motivation: The research team will effectively communicate with participants through regular check-ins, motivational messages, and feedback sessions.
5. Pilot Study: A pilot study will help identify potential barriers and refine strategies to enhance participant engagement early on.
6. Educational Support after the Study: In the final week, a nutritionist will conduct two nutritional education sessions for participants to support their post-study well-being. Participants will receive a personalized "Nutrition Card" with practical tips. These sessions are scheduled after the study to maintain dietary consistency during the 12-week intervention.
7. Community program: A community outreach program that will motivate and provide the conditions for participants to continue exercise training after the intervention ends.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older;
* Undergone breast cancer surgery with removal of at least one lymph node;
* Clinical diagnosis of stable unilateral breast cancer-related lymphedema;
* Willing and able to engage in exercise;
* Have not participated in a structured exercise program in the previous 6 months;
* Medical clearance to participate in the study.

Exclusion Criteria:

* Unstable lymphedema (therapist-delivered treatment and more than one arm infection requiring antibiotics in the past 3 months);
* Undergoing radiotherapy or chemotherapy by infusion for breast cancer;
* Bilateral lymphedema;
* Primary lymphedema;
* Uncontrolled heart disease (e.g., uncontrolled coronary heart disease, heart failure, uncontrolled hypertension);
* Type II diabetes;
* Psychological disorders (e.g., Alzheimer's, dementia, Parkinson's);
* Significant physical disabilities;
* Pregnancy and/or breastfeeding;
* Kidney disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 58 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Bioelectrical Impedance Spectroscopy - Lymphedema Index | 3 months
  To monitor tissue changes associated with BCRL, the ECW ratio will be assessed using BIS (Impedimed, SFB7, Pinkenba, Queensland, Australia). This method helps detect specific alterations in extracellular fluid containing lymph. Participants will be asked to lie down for 10 minutes, with their arms apart from their trunk, palms facing down, and legs apart, on a non-conductive surface. After cleaning the skin and removing all metals, electrodes will be placed on the hands and feet according to the manufacturer's instructions, aligning the sensing electrodes with the ulnar styloid and malleolus. Measurements will be taken on both the affected and unaffected upper limbs, and the Lymphedema Index (L-Dex) ratio will be calculated (unaffected limb impedance divided by the affected limb impedance). The L-Dex ratio is usually considered normal between -10.0 to 10.0. A score above 10.0 or an increase greater than 10 from baseline is indicative of potential BCRL.

SECONDARY OUTCOMES:
Range of motion | 3 months
  A goniometer will be used to assess active shoulder flexion and abduction with the participants in a standing position and the elbow fully extended. Each movement will be measured three times, and the average of these measurements will be calculated. Assessments will be conducted on both affected and unaffected upper limbs.
Anthropometric Measurements | 3 months
  Participants will be weighed wearing minimal clothing and no shoes. Height will be taken with a stadiometer (Seca, Hamburg, Germany) and following standardized procedures. Body mass index will be calculated by dividing weight (in kilograms) by the square of height (in meters).
Arm Circumferences | 3 months
  Arm circumferences of the affected and unaffected upper limbs will be measured with the arm positioned at 90° forward flexion using a soft tape measure, beginning at the midpoint of the ulna styloid ("0 cm" mark) and 10 cm intervals up to 40 cm proximal to the ulna styloid. Comparisons between affected and unaffected limbs will provide a quantitative assessment of lymphedema and allow for monitoring changes throughout the intervention.
Dual-energy X-ray Absorptiometry (DXA) | 3 months
  Participants will perform a whole-body DXA scan (Hologic Horizon DXA System, software QDR for Windows version 12.4, Waltham, USA) according to standardized procedures (ref). This equipment measures X-ray attenuation by pulsing between 70 and 140 kV in sync with the line frequency for each pixel in the scanned image. The same technician will position the participants, conduct the scan, and perform the analysis. DXA measurements will include whole-body and regional fat mass (FM) and fat-free mass (FFM). The same researcher will conduct all assessments and analysis to minimize inter-tester variation.
Dilution Techniques | 3 months
  Total body water (TBW) will be measured by deuterium oxide dilution using isotope ratio mass spectrometry. After an overnight fast, participants will provide a baseline urine sample, ingest 0.1 g/kg of 99.9% ²H₂O, and provide urine samples after equilibration for TBW determination.
  Extracellular water (ECW) will be assessed by sodium bromide (NaBr) dilution. Following a fast, participants will ingest 0.03 g/kg of 99% NaBr, and saliva samples will be collected after equilibration for analysis.
  Intracellular water (ICW) will be calculated as the difference between TBW and ECW.
Cardiopulmonary Exercise Test | 3 months
  A supervised incremental cardiopulmonary exercise test will be performed on a cycle ergometer. A 12-lead ECG and blood pressure will be monitored, and expired gases will be analyzed breath-by-breath using a calibrated portable gas analyzer. The protocol includes a 2-minute rest period, followed by stepwise workload increments until volitional exhaustion or clinical criteria are met. Peak oxygen consumption (VO₂peak) will be determined as the highest 20-second average during the final exercise stage, and recovery heart rate will be assessed at 60 and 120 seconds post-exercise.
Handgrip Strength | 3 months
  Upper body strength will be measured by maximal voluntary isometric contraction (MVIC) using a portable hand dynamometer. Participants will perform three 5-second maximal efforts with each hand in a standardized seated position, with 60 seconds of rest between trials. The best performance will be recorded as maximum voluntary isometric contraction.
The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 | 3 months
  The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30) will be administered to assess quality of life. The EORTC QLQ-C30 is a 30-item instrument designed to evaluate multiple dimensions of health, including five functional scales (physical, role, cognitive, emotional, and social functioning), three symptom scales (fatigue, pain, and nausea/vomiting), and a global health status/quality of life scale. It also includes items addressing cancer-related symptoms such as dyspnea, appetite loss, sleep disturbances, constipation, and diarrhea. The questionnaire uses a scoring methodology ranging from 0 to 100.
The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire BR23 | 3 months
  The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-BR23 (QLQ-BR23) will be administered to assess quality of life in breast cancer patients. The QLQ-BR23 is a complementary module to the QLQ-C30 and includes five multi-item domains evaluating body image, sexual functioning, systemic therapy side effects, and symptoms specific to the breast and arm. Scores are calculated using a 0-100 scale.
Disabilities of the Arm, Shoulder, and Hand | 3 months
  The Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire is a self-reported assessment tool comprising 30 items measuring upper extremity dysfunction's impact on daily activities. Each item is rated on a 5-point Likert scale, where one corresponds to no difficulty or interference, and 5 represents extreme difficulty or inability to perform the activity. A minimum of 27 completed items are required to calculate a score. The total score is determined by averaging the responses, subtracting one, and multiplying by 25 to yield a value out of 100. Higher DASH scores correspond to higher disability.
Hospital Anxiety and Depression Scale | 3 months
  The Hospital Anxiety and Depression Scale (HADS) will be used to evaluate depression and anxiety symptoms. This tool consists of 14 items divided into two seven-item subscales. Patients respond to each item using a four-point scale (graded 0 to 3), resulting in subscale scores ranging between 0 and 21. A score below 7 suggests no mood disorders, 8 to 10 suggests a possible mood disorder, and above 11 confirms the presence of mood disorders.
Physical Activity | 3 months
  Physical activity will be monitored using an ActiGraph GT3X accelerometer worn on the right hip for 7 consecutive days at baseline, week 6, and week 12. Data will be processed with ActiLife and GGIR software, with valid recordings defined as ≥10 hours/day on at least 2 weekdays and 1 weekend day. Outcomes will include time spent in different activity intensities and mean daily physical activity.
Hydration Status - Plasma osmolality | 3 months
  Blood samples will be collected to assess plasma osmolality (mOsm/L) using an osmometer (Mod OSMO1, Advanced Instruments, Canada) and plasma volume changes through hematocrit and hemoglobin measurements. The ion-selective method will determine Plasma sodium concentration (indirect ISE, Cobasc303 analyzer, Roche Diagnostics, UK). Blood samples will be collected from an antecubital vein through a ingle venipuncture and collected in tubes with EDTA, tubes with separating gel for the serum, and tubes with "heparin" for the plasma. The samples must be centrifuged for 10 minutes at 3000 rpm after retracting the clot to separate the serum. To obtain the plasma, they must be centrifuged immediately after collection for 10 minutes at 2000 rpm.
Hydration Status - Urine-Specific Gravity | 3 months
  A fasting baseline urine sample will be used to determine urine-specific gravity (USG) using a refractometer (PAL-10S, ATAGO, Japan).
Hydration Status - Hemoglobin | 3 months
  Hemoglobin will be quantified using the Beckman Coulter analyzer. Hemoglobin, obtained after erythrocyte lysis, is measured using absorption photometry. In this method, the blood is treated with a reagent that converts hemoglobin into a stable form, and the concentration is determined by absorbance at a specific wavelength. This method tracks hydration status and plasma volume shifts.
Hydration Status - Hematocrit | 3 months
  Hematocrit will be quantified using the Beckman Coulter analyzer. Hematocrit (Hct) is determined indirectly from the red blood cell count (RBC) and mean corpuscular volume (MCV) using the formula Hct = (RBC × MCV) / 10. This method tracks hydration status and plasma volume shifts.
Ultrassound Assessment | 3 months
  Acute muscular and fluid responses to exercise will be assessed at baseline, week 6, and week 12. Ultrasound imaging (12-MHz linear probe) will be used to measure biceps brachialis thickness before and after a training session. Measurements will be taken at a standardized anatomical site on the upper arm, with images analyzed using ImageJ software to determine muscle thickness between superficial and deep fascia. The same trained assessor will perform all scans to ensure consistency.
  Percentage changes in muscle thickness across time points will be calculated and interpreted alongside plasma volume assessments (hematocrit-based), providing insight into fluid shifts and acute muscular responses to training.
Inflammatory Profile - Creatine Kinase | 3 months
  A qualified phlebotomist will collect Venous blood samples from the unaffected arm. After the biological samples have been separated, creatine kinase (CK) will be measured using the enzymatic-UV and immunoturbidimetric methods on the Cobas c303 analyzer.
Inflammatory Profile - C-reactive Protein | 3 months
  A qualified phlebotomist will collect Venous blood samples from the unaffected arm. After the biological samples have been separated, c-reactive protein (CRP) will be measured using the enzymatic-UV and immunoturbidimetric methods on the Cobas c303 analyzer.
Inflammatory Profile - Interleukin-6 | 3 months
  A qualified phlebotomist will collect Venous blood samples from the unaffected arm. After the biological samples have been separated, Interleukin-6 (IL-6) will be quantified using the electrochemiluminescence method (ECLIA, Cobas e411 analyzer, Roche Diagnostics, UK).
Habitual Dietary Intake | 3 months
  A trained nutritionist will conduct three non-consecutive 24-hour dietary recalls (including one weekend day) to estimate dietary intake. The multiple pass method - a five-step approach designed to enhance the complete and accurate registration of all foods and beverages consumed, including amount (portion size), brand (if relevant), and preparation (e.g., cooking methods) over 24 hours - will be used. The food portions will be quantified using visual aids depicting various portion sizes. Data from the records will be inserted into Food Processor Plus® (version 10.12.0.0, ESHA Research, USA) for analysis. Mean total energy, macro- and micronutrients, and fluid intake will be calculated by averaging all recall days.

CONTACTS AND LOCATIONS:
Overall Officials: Rúben Francisco, PhD, Principal Investigator — Polytechnic Institute of Rio Maior
Locations (1):
- Faculdade de Motricidade Humana, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No